CLINICAL TRIAL: NCT05450458
Title: Safety and Effectiveness of Hyaluronic Acid and Sorbitol With Overuse Knee Pain in Sportsmen
Brief Title: Hyaluronic Acid in Overuse Knee Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Regional Tlalnepantla (Other Government)
Responsible Party: Principal Investigator, Julio Carlos Velez de Lachica, Head of orthopedic surgery department, Hospital Regional Tlalnepantla
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEI/0504/PI/2022
Record Dates: First submitted 2022-06-17; First posted 2022-07-08 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Overuse Injury; Body Mass Index in Athletes
Keywords: KNEE; PAIN; SPORTSMEN; HYALURONIC ACID
MeSH Terms: conditions — Cumulative Trauma Disorders; Pain | interventions — Hyaluronic Acid; Viscosupplementation

STUDY DESIGN:
Intervention Model Description: A study group will be integrated which will be evaluated before the intervention and after 15 days, 3 and 6 subsequent months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyaluronic Acid group (Experimental): All overuse knee syndrome participants after both knee joint infiltration with two doses each of Synolis VA (2ml = 40 milligrams of hyaluronic acid with 80 milligrams of sorbitol).
  Interventions: Drug: KNEE JOINT INFILTRATION WITH HYALURONIC ACID WITH SORBITOL SYNOLIS VA

INTERVENTIONS:
Drug: KNEE JOINT INFILTRATION WITH HYALURONIC ACID WITH SORBITOL SYNOLIS VA — KNEE INFILTRATION WITH HYALURONIC ACID WITH SORBITOL IN SPORTSMEN
  Other Names: VISCOSUPPLEMENTATION WITH SYNOLIS VA

SUMMARY:
Sports activity represents part of day living people, a knee pain originated by high demand joint activity could represent a limitation to continue sports. The aim of this clinical trial is demonstrate the effects of hyaluronic acid in sportsmen with knee pain.

DETAILED DESCRIPTION:
Sports activities have become a fundamental part of our daily life, this has led to an overuse of load joints, being the knee the most relevant. Overuse injuries of the knee result from microtrauma associated with physical activity and exercise that exceeds the strength of the cartilage tissue.

The purpose of this study is to evaluate the usefulness and safety of hyaluronic acid in athlete patients with knee overuse syndrome. Investigators hypothesis is that hyaluronic acid y safe and can improve symptoms of knee pain in sports patients. . Scores recorder data will be made at 15 days, then at 3 and 6 months after two knee injections of hyaluronic acid with sorbitol (Synolis VA).

Synolis VA is a viscoelastic, sterile, non-pyrogenic, isotonic, buffered solution of 2% hyaluronic acid. The hyaluronic acid used in synolis VA is obtained from bacterial fermentation and has a high molecular weight of 2 mdaltons, it has a neutral pH of 6.8 - 7.4 like synovial fluid. High concentration and high molecular weight of hyaluronic acid combined with sorbitol limits its degradation and confers the capacity of viscoelastic solution to restore joint lubrication and shock absorption properties.

This research protocol has been approve by the ethics and research Institutional committee in ISSEMyM Tlalnepantla Estado de Mexico number: CEI/0504/PI./2022. All participants must sign a informed consent to confirm be part fo this study.

ELIGIBILITY:
Inclusion Criteria:

* - Patients with knee pain for more than 3 months
* Patients between 30 and 55 years old
* Patients without a history of previous knee joint surgery.
* Patients without chronic-degenerative diseases such as diabetes, hypertension, rheumatoid arthritis or other autoimmune diseases.
* Patients who perform impact social sports at least 3 times a week for more than 1 hour in the last 3 months prior to treatment.
* Patients without a history of allergies to non-steroidal anti-inflammatory drugs.
* Patients with no history of infection in or around the knee.

Exclusion Criteria:

* - Patients who cannot be categorized as social athletes.
* Patients with an associated sports injury that limits their sports practice.
* Patients who have a treatment associated with knee pain independent of that established in the study protocol.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Issemym Tlalnepantla, Tlanepantla, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel DR, Villalobos A. Evaluation and management of knee pain in young athletes: overuse injuries of the knee. Transl Pediatr. 2017 Jul;6(3):190-198. doi: 10.21037/tp.2017.04.05. PMID 28795010
- [Background] Nicolini AP, de Carvalho RT, Matsuda MM, Sayum JF, Cohen M. Common injuries in athletes' knee: experience of a specialized center. Acta Ortop Bras. 2014;22(3):127-31. doi: 10.1590/1413-78522014220300475. PMID 25061417
- [Background] Fuller CW, Ekstrand J, Junge A, Andersen TE, Bahr R, Dvorak J, Hagglund M, McCrory P, Meeuwisse WH. Consensus statement on injury definitions and data collection procedures in studies of football (soccer) injuries. Br J Sports Med. 2006 Mar;40(3):193-201. doi: 10.1136/bjsm.2005.025270. PMID 16505073
- [Background] Majewski M, Susanne H, Klaus S. Epidemiology of athletic knee injuries: A 10-year study. Knee. 2006 Jun;13(3):184-8. doi: 10.1016/j.knee.2006.01.005. Epub 2006 Apr 17. PMID 16603363
- [Background] Wilder RP, Sethi S. Overuse injuries: tendinopathies, stress fractures, compartment syndrome, and shin splints. Clin Sports Med. 2004 Jan;23(1):55-81, vi. doi: 10.1016/S0278-5919(03)00085-1. PMID 15062584
- [Background] Aicale R, Tarantino D, Maffulli N. Overuse injuries in sport: a comprehensive overview. J Orthop Surg Res. 2018 Dec 5;13(1):309. doi: 10.1186/s13018-018-1017-5. PMID 30518382
- [Background] Paoloni M, Bernetti A, Belelli A, Brignoli O, Buoso S, Caputi AP, Catani F, Coclite D, Fini M, Mantovani L, Migliore A, Napoletano A, Viora U, Santilli V. Appropriateness of clinical and organizational criteria for intra-articular injection therapies in osteoarthritis. A Delphi method consensus initiative among experts in Italy. Ann Ist Super Sanita. 2015;51(2):131-8. doi: 10.4415/ANN_15_02_11. PMID 26156184
- [Background] Yang J, Tibbetts AS, Covassin T, Cheng G, Nayar S, Heiden E. Epidemiology of overuse and acute injuries among competitive collegiate athletes. J Athl Train. 2012 Mar-Apr;47(2):198-204. doi: 10.4085/1062-6050-47.2.198. PMID 22488286
- [Background] Drawer S, Fuller CW. Propensity for osteoarthritis and lower limb joint pain in retired professional soccer players. Br J Sports Med. 2001 Dec;35(6):402-8. doi: 10.1136/bjsm.35.6.402. PMID 11726474
- [Background] Vannini F, Spalding T, Andriolo L, Berruto M, Denti M, Espregueira-Mendes J, Menetrey J, Peretti GM, Seil R, Filardo G. Sport and early osteoarthritis: the role of sport in aetiology, progression and treatment of knee osteoarthritis. Knee Surg Sports Traumatol Arthrosc. 2016 Jun;24(6):1786-96. doi: 10.1007/s00167-016-4090-5. Epub 2016 Apr 4. PMID 27043343
- [Background] Frohlich S, Pazeller S, Cherati AS, Muller E, Frey WO, Sporri J. Overuse injuries in the knee, back and hip of top elite female alpine skiers during the off-season preparation period: prevalence, severity and their association with traumatic preinjuries and training load. BMJ Open Sport Exerc Med. 2020 Dec 24;6(1):e000892. doi: 10.1136/bmjsem-2020-000892. eCollection 2020. PMID 33408876
- [Background] Rincon GA, Vyas D, Zhou J, Fu FH, Oiestad BE, Holm I, Aune AK, Gunderson R, Myklebust G, Engebretsen L, Fosdahl M, Risberg MA. "Knee function and prevalence of knee osteoarthritis after anterior cruciate ligament reconstruction: a prospective study with 10 to 15 years of follow-up". Letter to the editor. Am J Sports Med. 2011 Apr;39(4):NP3; author reply NP3-4. doi: 10.1177/0363546511403704. No abstract available. PMID 21460071
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of osteo-arthrosis. Ann Rheum Dis. 1957 Dec;16(4):494-502. doi: 10.1136/ard.16.4.494. No abstract available. PMID 13498604
- [Background] Hunter DJ, Lo GH, Gale D, Grainger AJ, Guermazi A, Conaghan PG. The reliability of a new scoring system for knee osteoarthritis MRI and the validity of bone marrow lesion assessment: BLOKS (Boston Leeds Osteoarthritis Knee Score). Ann Rheum Dis. 2008 Feb;67(2):206-11. doi: 10.1136/ard.2006.066183. Epub 2007 May 1. PMID 17472995
- [Background] Maffulli N, Regine R, Carrillo F, Minelli S, Beaconsfield T. Ultrasonographic scan in knee pain in athletes. Br J Sports Med. 1992 Jun;26(2):93-6. doi: 10.1136/bjsm.26.2.93. PMID 1623366
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] Luyten FP, Denti M, Filardo G, Kon E, Engebretsen L. Definition and classification of early osteoarthritis of the knee. Knee Surg Sports Traumatol Arthrosc. 2012 Mar;20(3):401-6. doi: 10.1007/s00167-011-1743-2. Epub 2011 Nov 8. PMID 22068268
- [Background] Hoemann C, Kandel R, Roberts S, Saris DB, Creemers L, Mainil-Varlet P, Methot S, Hollander AP, Buschmann MD. International Cartilage Repair Society (ICRS) Recommended Guidelines for Histological Endpoints for Cartilage Repair Studies in Animal Models and Clinical Trials. Cartilage. 2011 Apr;2(2):153-72. doi: 10.1177/1947603510397535. PMID 26069577
- [Background] Peterfy CG, Guermazi A, Zaim S, Tirman PF, Miaux Y, White D, Kothari M, Lu Y, Fye K, Zhao S, Genant HK. Whole-Organ Magnetic Resonance Imaging Score (WORMS) of the knee in osteoarthritis. Osteoarthritis Cartilage. 2004 Mar;12(3):177-90. doi: 10.1016/j.joca.2003.11.003. PMID 14972335
- [Background] Leslie M. Knee osteoarthritis management therapies. Pain Manag Nurs. 2000 Jun;1(2):51-7. doi: 10.1053/jpmn.2000.7782. PMID 11706459
- [Background] Demange MK, Sisto M, Rodeo S. Future trends for unicompartmental arthritis of the knee: injectables & stem cells. Clin Sports Med. 2014 Jan;33(1):161-74. doi: 10.1016/j.csm.2013.06.006. Epub 2013 Jul 19. PMID 24274853
- [Background] Sandmark H, Hogstedt C, Lewold S, Vingard E. Osteoarthrosis of the knee in men and women in association with overweight, smoking, and hormone therapy. Ann Rheum Dis. 1999 Mar;58(3):151-5. doi: 10.1136/ard.58.3.151. PMID 10364912
- [Background] Fransen M, McConnell S. Land-based exercise for osteoarthritis of the knee: a metaanalysis of randomized controlled trials. J Rheumatol. 2009 Jun;36(6):1109-17. doi: 10.3899/jrheum.090058. Epub 2009 May 15. PMID 19447940
- [Background] de Sire A, Agostini F, Lippi L, Mangone M, Marchese S, Cisari C, Bernetti A, Invernizzi M. Oxygen-Ozone Therapy in the Rehabilitation Field: State of the Art on Mechanisms of Action, Safety and Effectiveness in Patients with Musculoskeletal Disorders. Biomolecules. 2021 Feb 26;11(3):356. doi: 10.3390/biom11030356. PMID 33652804
- [Background] Hiemstra LA, Kerslake S, Irving C. Anterior knee pain in the athlete. Clin Sports Med. 2014 Jul;33(3):437-59. doi: 10.1016/j.csm.2014.03.010. Epub 2014 May 24. PMID 24993409
- [Background] Brophy RH, Fillingham YA. AAOS Clinical Practice Guideline Summary: Management of Osteoarthritis of the Knee (Nonarthroplasty), Third Edition. J Am Acad Orthop Surg. 2022 May 1;30(9):e721-e729. doi: 10.5435/JAAOS-D-21-01233. PMID 35383651
- [Background] Trojian TH, Concoff AL, Joy SM, Hatzenbuehler JR, Saulsberry WJ, Coleman CI. AMSSM Scientific Statement Concerning Viscosupplementation Injections for Knee Osteoarthritis: Importance for Individual Patient Outcomes. Clin J Sport Med. 2016 Jan;26(1):1-11. doi: 10.1097/JSM.0000000000000274. PMID 26562453
- [Background] Kalkhoven J, Coutts AJ, Impellizzeri FM. 'Training load error' is not a more accurate term than 'overuse' injury. Br J Sports Med. 2020 Aug;54(15):934-935. doi: 10.1136/bjsports-2019-101710. Epub 2020 Feb 24. No abstract available. PMID 32094146
- [Background] Odole AC, Agbomeji OT, Onyeso OKK, Ojo JO, Odunaiya NA. Perspectives of Nigerian Athletes About Physiotherapy Services in Sports Injury Management: Implications for Rehabilitation. J Sport Rehabil. 2021 Feb 16;30(6):876-883. doi: 10.1123/jsr.2020-0292. PMID 33596541
- [Background] Ammar TY, Pereira TA, Mistura SL, Kuhn A, Saggin JI, Lopes Junior OV. Viscosupplementation for treating knee osteoarthrosis: review of the literature. Rev Bras Ortop. 2015 Aug 5;50(5):489-94. doi: 10.1016/j.rboe.2015.07.007. eCollection 2015 Sep-Oct. PMID 26535192
- [Background] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Background] Higgins LD, Taylor MK, Park D, Ghodadra N, Marchant M, Pietrobon R, Cook C; International Knee Documentation Committee. Reliability and validity of the International Knee Documentation Committee (IKDC) Subjective Knee Form. Joint Bone Spine. 2007 Dec;74(6):594-9. doi: 10.1016/j.jbspin.2007.01.036. Epub 2007 Aug 6. PMID 17888709
- [Background] Kujala UM, Kaprio J, Sarna S. Osteoarthritis of weight bearing joints of lower limbs in former elite male athletes. BMJ. 1994 Jan 22;308(6923):231-4. doi: 10.1136/bmj.308.6923.231. PMID 8111258
- [Background] Emanuel EJ, Wendler D, Grady C. What makes clinical research ethical? JAMA. 2000 May 24-31;283(20):2701-11. doi: 10.1001/jama.283.20.2701. PMID 10819955
- See also: Tiu T, Craig Van Dien MD. Knee overuse disorders — https://now.aapmr.org/knee-overuse-disorders/

RESULTS

PARTICIPANT FLOW:
Groups:
- Athletes With Overuse Knee Syndrome: Patients who are considered athletes of moderate or high impact activities are those who practice a sport of this type at least 3 times per week for at least 1 hour, and who also experience knee pain related to the sports activity..
Period: Overall Study
Arm/Group | Athletes With Overuse Knee Syndrome
Started | 64
Completed | 60
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Groups:
- Athletes With Overuse Knee Syndrome: Patients who are considered athletes of moderate or high impact activities are those who practice a sport of this type at least 3 times per week for at least 1 hour, and who also experience knee pain related to the sports activity. The diagnosis was based on clinical evaluation, ultrasound, and X-ray findings. Eligibility criteria included patients aged 30 to 55 years who participate in moderate to high-impact knee sports activities at least three times per week, with a minimum duration of one hour per session; absence of surgical intervention, ligament or meniscal injuries, acute or chronic infections, or sequelae injuries in the pelvic limbs; ability to complete the 6-month follow-up without the use of NSAIDs and full adherence to the study protocol. All participants were treated with two HA-Sorbitol knee injections by the same technique and surgeon and evaluated with the KOOS and IKDC scores over time at baseline, 15 days, 3 months and 6 months.
Arm/Group | Athletes With Overuse Knee Syndrome
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants] — Athletes diagnosed with knee overuse syndrome were recruited, undergoing a thorough physical exam and ultrasound to rule out ligament, osteochondral, or meniscal injuries. Results of the IKDC scale (International Knee Documentation Committee) and the KOOS scale (Knee injury and Osteoarthritis Outcome Score) were collected over time.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 60
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 60
IKDC baseline [Mean (Standard Deviation); unit: percentage] — This score is derived from the patient's responses in the IKDC scale (International Knee Documentation Committee) measures knee function with a scoring range from 0 to 87, where 87 represents 100% function (best possible outcome) and 0 represents the worst function. In this study, results are presented as percentages rather than raw score points
  percentage | 65 (10.6)
KOOS baseline [Mean (Standard Deviation); unit: percentage] — The KOOS scale (Knee injury and Osteoarthritis Outcome Score) is used to assess knee-related quality of life, symptoms, pain, activities of daily living, and sport/recreation function, with scores ranging from 0 to 100, where higher scores indicate better knee health.
  percentage | 68 (10.6)
BMI [Mean (Standard Deviation); unit: kg/m²] — body mass index at baseline
  kg/m² | 24 (3.18)
Primary sport [Count of Participants; unit: Participants] — It is defined as the high-level or high-impact sport that the participant engaged in.
  Participants
    running | 16
    tennis | 12
    hiit | 3
    aerobics | 2
    grit | 4
    weight lifting | 4
    crossfit | 9
    montain biker | 1
    soccer | 6
    jazz dancer | 3
Athlete type [Count of Participants; unit: Participants] — If the participant practice a Social, Amateur or Professional sport activity
  Participants
    SOCIAL | 12
    AMATEUR | 38
    PROFESSIONAL | 10

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Hyaluronic Acid With Sorbitol (SYNOLIS VA) in Overuse Knee Syndrome Assessed With the Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: To demonstrate that two doses of intra-articular injection of Synolis VA® for the overuse knee syndrome in sportsmen decrease the pain during spots and day-living activities by measured the improvement of knee symptoms through the KOOS score:
  - The Knee injury and Osteoarthritis Outcome Score: Evaluate Symptoms + Stiffness subtotal, Pain, Function, daily living, sports and recreational activities and quality of life. Each variable has a percentage score from 0 to 100%, at the end the results are averaged, obtaining a final percentage where 100% means a healthy knee with out discomfort. As the percentage approaches 0%, the severity of knee discomfort or injury increases.
Time Frame: Baseline, 15 days, 3 months, and 6 months
Population: 60 athletes diagnosed with overuse knee syndrome due to sports were included. Synolis VA was applied as a treatment, and participants were evaluated over time using the KOOS (Knee injury and Osteoarthritis Outcome Score) at basal, 15 days, 3 months and 6 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- KOOS Score: All overuse knee syndrome participants after both knee joint infiltration with two doses each of Synolis VA (2ml = 40 milligrams of hyaluronic acid with 80 milligrams of sorbitol). Assessed over time with the KOOS score.
Arm/Group | KOOS Score
Number analyzed (Participants) | 60
score on a scale
  KOOS Basal | 68 (10.6)
  KOOS 15 days | 78 (8.27)
  KOOS 3 Months | 84 (8.78)
  KOOS 6 Months | 88 (7.63)
Statistical Analysis 1: Comparison: KOOS Score; The statistical analysis will use the Friedman test, as the Shapiro-Wilk test confirmed a non-normal distribution. Conover's post hoc test with Bonferroni correction will adjust for multiple comparisons. The null hypothesis states that hyaluronic acid injections with sorbitol do not significantly improve KOOS function and pain scores over time. A power analysis was performed to ensure an adequate sample size for detecting clinically meaningful differences; Test type: Other — This study assessed longitudinal effects within a single patient group. Statistical power was calculated using a significance level of 0.05, 80% power, and 60 patients, accounting for KOOS score variability over time. The Friedman test was applied with post hoc analyses (Conover and Bonferroni). Since treatments were not compared, no non-inferiority or equivalence margin was defined; p < 0.001, Friedman Test — P-values were adjusted for multiple comparisons using the Bonferroni method, and the a priori threshold for statistical significance was set at 0.05; Post hoc pairwise comparisons were adjusted using the Bonferroni method, and the a priori significance level was set at 0.05; Median Change Baseline to month 6 = 0.22, 95% CI 2-sided [0.15 to 0.23] — The value represents the intra-individual median KOOS improvement from baseline to month 6 after treatment. Changes were evaluated across time points within a single cohort

2. Primary Outcome: Efficacy of Hyaluronic Acid With Sorbitol (SYNOLIS VA) in Overuse Knee Syndrome Assessed With the International Knee Documentation Committee Score (IKDC)
Description: To evaluate the effectiveness of two intra-articular injections of Synolis VA in improving knee functionality in athletes with overuse knee syndrome, the International Knee Documentation Committee (IKDC) Scale was used. This validated tool assesses knee function, symptoms, and the ability to perform sports-related activities. It consists of individual items evaluating pain, stiffness, swelling, instability, daily physical function, and athletic performance. While the scale's raw score ranges from 0 to 87, results are converted into a percentage format, where 87 corresponds to 100% functional capacity-the best possible knee function-and 0 represents the worst condition."
Time Frame: Baseline, 15 days, 3 months, and 6 months
Population: IKDC score was collected from 60 participants after the knee injection with two doses of synolis VA, basal, 15 days, 3 months and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- IKDC SCORE: All overuse knee syndrome participants after both knee joint infiltration with two doses each of Synolis VA (2ml = 40 milligrams of hyaluronic acid with 80 milligrams of sorbitol). Assessed over time with the IKDC score.
Arm/Group | IKDC SCORE
Number analyzed (Participants) | 60
score on a scale
  IKDC basal | 65 (10.60)
  IKDC 15 DAYS | 74 (11.05)
  IKDC 3 MONTHS | 81 (8.91)
  IKDC 6 MONTHS | 83 (8.88)
Statistical Analysis 1: Comparison: IKDC SCORE; The statistical analysis will use the Friedman test, as the Shapiro-Wilk test confirmed a non-normal distribution. Conover's post hoc test with Bonferroni correction will adjust for multiple comparisons. The null hypothesis states that hyaluronic acid injections with sorbitol do not significantly improve IKDC function and pain scores over time. A power analysis was performed to ensure an adequate sample size for detecting clinically meaningful differences; Test type: Other — This study assessed longitudinal effects within a single patient group. Statistical power was calculated using a significance level of 0.05, 80% power, and 60 patients, accounting for IKDC score variability over time. The Friedman test was applied with post hoc analyses (Conover and Bonferroni). Since treatments were not compared, no non-inferiority or equivalence margin was defined; p = 0.01, Friedman Test — [p-value comment as in outcome 1, analysis 1]; The overall p-value is unadjusted. The a priori significance level was set at 0.05 to robustly control the Type I error; Median Baseline to Month 6 = 0.18, 95% CI 2-sided [0.12 to 0.24] — This value represents the intra-individual median IKDC improvement from baseline to 6 months after treatment. The analysis was conducted within a single cohort without comparator arms

3. Secondary Outcome: Safety of Hyaluronic Acid With Sorbitol (SYNOLIS VA ®) in Overuse Knee Syndrome by the Number of Adverse Effects in Participants.
Description: Evaluate the SYNOLIS VA ® safety after two doses of intra articular injection by tracking the number of patient withdrawals and their adverse events including: skin irritation, knee redness, local pain for more than 24 hours, edema for more than 48 hours and itching at the application site.
Time Frame: 6 months
Population: Sixty patients were evaluated after receiving two doses of Synolis VA per knee. Assessments were performed at baseline, 15 days, 3 months, and 6 months.
Measure: Count of Participants; unit: Participants
Groups:
- Athletes With Overuse Knee Syndrome: Patients who are considered athletes of moderate or high impact activities are those who practice a sport of this type at least 3 times per week for at least 1 hour, and who also experience knee pain related to the sports activity. Sixty patients were evaluated after receiving two doses of Synolis VA per knee. Assessments were performed at baseline, 15 days, 3 months, and 6 months. No adverse events were observed in any case.
Arm/Group | Athletes With Overuse Knee Syndrome
Number analyzed (Participants) | 60
Participants | 0

4. Secondary Outcome: Six-Month Functional Improvement in Knee Function (IKDC and KOOS) in Athletes With Overuse Knee Syndrome With Elevated BMI Following Synolis VA Injections
Description: This measure evaluates the change in knee function over a six-month period in athletes with an elevated body mass index (BMI > 25) diagnosed with overuse knee syndrome and treated with intra-articular injections of Synolis VA®. Two validated patient-reported outcome instruments are used: the International Knee Documentation Committee Subjective Knee Evaluation Form (scale: 0 = poorest function, 100 = best function) and the Knee Injury and Osteoarthritis Outcome Score (scale: 0 = worst outcome, 100 = best outcome). Higher scores indicate better knee functionality. Baseline scores are compared with six-month scores to assess functional improvement.
Time Frame: 6 months post-treatment
Population: Analysis includes 22 athletes with a BMI >25 who had complete baseline and six-month data for both the International Knee Documentation Committee Subjective Knee Evaluation Form and the Knee Injury and Osteoarthritis Outcome Score. Normality was assessed using the Shapiro-Wilk test, and since the data were non-normally distributed, paired comparisons were made using the Wilcoxon Signed-Rank Test
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- BMI Elevated IKDC Score: Athletes with an elevated body mass index (BMI > 25) who have been diagnosed with overuse knee syndrome and are treated with two intra-articular injections of Synolis VA. Participants in this group are assessed at baseline and again at six months using the International Knee Documentation Committee Scale (IKDC) to evaluate changes in knee functionality over time
- BMI Elevated KOOS Score: Athletes with an elevated body mass index (BMI > 25) who have been diagnosed with overuse knee syndrome and are treated with two intra-articular injections of Synolis VA. Participants in this group are assessed at baseline and again at six months using the Knee injury and Osteoarthritis Outcome Score (KOOS) to evaluate changes over knee related quality of life, symptoms, pain, activities of daily living, and sport/recreation function over time.
Arm/Group | BMI Elevated IKDC Score | BMI Elevated KOOS Score
Number analyzed (Participants) | 22 | 22
score on a scale | 83.1 [79.9 to 86.1] | 85 [81 to 91]
Statistical Analysis 1: Comparison: BMI Elevated IKDC Score; The analysis was conducted under the null hypothesis of no change in knee function across time. Data normality was assessed using the Shapiro-Wilk test. Changes across the four time points (baseline, 15 days, 3 months, and 6 months) were evaluated using the Friedman test. Pairwise comparisons were performed post hoc using the Wilcoxon Signed-Rank Test with Bonferroni correction at a 5% significance threshold; Test type: Superiority — This is a superiority analysis. Data normality was first assessed with the Shapiro-Wilk test, and due to non-normal distributions, a Wilcoxon Signed-Rank Test was applied to compare paired baseline and six-month IKDC score; p = 0.001, Wilcoxon Signed-Rank Test — P-values from pairwise comparisons were adjusted using the Bonferroni method to control for multiple testing. The global p-value from the Friedman test was not adjusted. An a priori threshold for statistical significance was set at p < 0.05; Friedman test conducted with 3 degrees of freedom. Bonferroni correction applied in pairwise Wilcoxon post hoc comparisons; Baseline to month 6 = 0.18, 95% CI 2-sided [0.14 to 0.21] — Median IKDC improvement from baseline to 6 months in 22 athletes with elevated BMI (≥25). No comparator group was used. Confidence interval calculated via bootstrap (resampling with 1,000 iterations)
Statistical Analysis 2: Comparison: BMI Elevated KOOS Score; The analysis was conducted under the null hypothesis of no change in knee function between baseline and six months. The study was designed with sufficient power to detect clinically meaningful improvements, with significance determined at a conventional level; Test type: Superiority — This is a superiority analysis. Data normality was first assessed with the Shapiro-Wilk test, and due to non-normal distributions, a Wilcoxon Signed-Rank Test was applied to compare paired baseline and six-month KOOS score; p < 0.001, Wilcoxon Signed-Rank Test — The p-values reported were not adjusted for multiple comparisons, and the a priori threshold for statistical significance was set at p < 0.05; [statistical method as in outcome 4, analysis 1]; Baseline to Month 6 = 18.5, 95% CI 2-sided [13 to 22] — Median KOOS improvement from baseline to 6 months in 22 athletes with elevated BMI. CI calculated via bootstrap resampling (1,000 iterations). No comparator group was involved

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 6-month intervention period for each participant.
Description: The collection included active surveillance for predefined adverse events of interest: skin erythema, joint effusion, localized inflammation, pain, pyrexia (≥38°C), joint infection, and functional impairment after knee injection.
Arm/Group | Athletes With Overuse Knee Syndrome
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT05450458/Prot_SAP_ICF_000.pdf